CLINICAL TRIAL: NCT06417775
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Ubrogepant for the Preventive Treatment of Menstrual Migraine With an Open-Label Extension
Brief Title: Study of Oral Ubrogepant to Assess Adverse Events and Change in Disease Activity in Adult Participants With Menstrual Migraine
Acronym: UBRO MM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M23-714
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Migraine
Keywords: Migraine; Menstrual Migraine; Ubrogepant; UBRELVY
MeSH Terms: conditions — Migraine Disorders | interventions — ubrogepant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Double-Blind Period: Ubrogepant (Experimental): Participants will receive ubrogepant during the double-blind period.
  Interventions: Drug: Ubrogepant
- Double-Blind Period: Placebo for Ubrogepant (Experimental): Participants will receive placebo during the double-blind period.
  Interventions: Drug: Placebo for Ubrogepant
- Open-Label Extension Period: Ubrogepant (Experimental): Eligible participants from Double-Blind period may continue to receive ubrogepant during the open-label extension period.
  Interventions: Drug: Ubrogepant

INTERVENTIONS:
Drug: Ubrogepant — Oral Tablets
  Other Names: UBRELVY
  Arms: Double-Blind Period: Ubrogepant; Open-Label Extension Period: Ubrogepant
Drug: Placebo for Ubrogepant — Oral Tablets
  Arms: Double-Blind Period: Placebo for Ubrogepant

SUMMARY:
A migraine is a moderate to severe headache typically on one side of the head. A migraine attack is a headache that may be accompanied by throbbing, nausea, vomiting, sensitivity to light and sound, or other symptoms. Menstrual migraine (MM) is defined as migraine attacks that occur within the perimenstrual period (PMP) in at least 2 out of 3 menstrual cycles. The PMP is from 2 days before the onset of menstrual bleeding to 2 days after. This study will assess how safe and effective ubrogepant is in treating menstrual migraine. Adverse Events and change in disease activity will be assessed.

Ubrogepant is an investigational drug being developed for short-term prevention of menstrual migraine. Participants will be randomly assigned to one of the 2 groups to receive either ubrogepant or placebo. Around 496 adult female participants with menstrual migraine will be enrolled in approximately 100 sites in the United States and Puerto Rico.

Participants will receive oral ubrogepant tablets once daily for 7 consecutive days starting 3 days prior to estimated onset of menses per cycle for 3 PMPs during double-blind period (16 weeks). Eligible participants may continue to receive oral ubrogepant tablets once daily for 7 consecutive days per cycle starting 3 days prior to estimated onset of menses during open-label extension period (52 weeks).

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will collect data daily in electronic diaries and attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* At least a 1-year history of migraine with or without aura.
* Have experienced migraine attacks in at least 2 of 3 perimenstrual periods (PMPs) during the screening period.
* Collection of daily eDiary data for 3 perimenstrual periods during the up to 16-week screening period to confirm a menstrual migraine (MM) diagnosis.
* Have regular menstrual cycles of between 21-35 days in length.
* Less than 15 headache days per month.
* At least 70% compliance completing screening period and at least 3 out of 5 days of ediary data in each of 3 screening PMP.

Exclusion Criteria:

* History of migraine with brainstem aura, hemiplegic migraine, or retinal migraine.
* Clinically significant history of cardiovascular or cerebrovascular disease per the investigator's opinion.
* Clinically significant abnormalities in the physical examination as determined by the investigator.
* Clinically significant hematologic, endocrine, pulmonary, renal, hepatic, gastrointestinal, gynecological, or neurologic disease per the investigator's opinion.
* Acute headache medication overuse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Number of Migraine Days Occurring During Perimenstrual Periods (PMPs) Across the Double-Blind Treatment Period | Up to approximately 16 Weeks
  A migraine day is defined as any calendar day on which a headache occurs which meets criteria listed in the protocol as per eDiary.
Number of Participants With Adverse Events (AEs) | Up to approximately 68 Weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change From Baseline in Number of Headache Days Occurring During Perimenstrual Periods (PMPs) Across the Double-Blind Treatment Period | Up to approximately 16 Weeks
  A headache day is defined as any calendar day on which headache pain lasting 2 hours or longer occurs unless an acute headache medication was used after the start of the headache, in which case no minimum duration will be specified.
Change From Baseline in Number of Moderate or Severe Headache Days During Perimenstrual Periods (PMPs) Across the Double-Blind Treatment Period | Up to approximately 16 Weeks
  A headache day is defined as any calendar day on which headache pain lasting 2 hours or longer occurs unless an acute headache medication was used after the start of the headache, in which case no minimum duration will be specified.
Change From Baseline in Number of Migraine Days With Moderate or Severe Headache During Perimenstrual Periods (PMPs) Across the Double-Blind Treatment Period | Up to approximately 16 Weeks
  A migraine day is defined as any calendar day on which a headache occurs which meets criteria listed in the protocol as per eDiary.
Percentage of Participants With No Disability/ Mild Impairment for most (>= 65%) of PMP Days | Up to approximately 16 Weeks
  Functional Disability Scale (FDS) is a single item used to measure the participant's level of functional disability. Participants will be asked to rate the performance of daily activities in the past 24 hours using 4 response options ranging from "No disability, able to function normally" to "Severely impaired, cannot do all or most things, bed rest may be necessary."
Change From Baseline in Acute Medication Use Days During the Perimenstrual Periods (PMPs) Across the Double-Blind Treatment Period | Up to approximately 16 Weeks
  An acute medication use day is defined as any day on which a participant reports, per eDiary, the intake of allowed medication(s) for the acute treatment of migraine.
Percentage of Participants Achieving >= 50% Reduction in Number of Migraine Days During the Perimenstrual Periods (PMPs) Across the Double-Blind Treatment Period | Up to approximately 16 Weeks
  A migraine day is defined as any calendar day on which a headache occurs which meets criteria listed in the protocol as per eDiary.
Percentage of Participants Achieving "Not at all limited" or "A little limited" Daily Activity Level for Most (>= 65%) of PMP Days | Up to approximately 16 Weeks
  Activity Level is a single-item used to assess overall limitations with performing daily activities over 24 hours with a 5-level response ranging from "Not at all limited" to "Unable to do daily activities."

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (106):
- United States (103):
  - Central Research Associates /ID# 260161, Birmingham, Alabama
  - Rehabilitation & Neurological Services /ID# 275593, Huntsville, Alabama
  - MD First Research - Chandler /ID# 262564, Chandler, Arizona
  - Gilbert Neurology /ID# 260179, Gilbert, Arizona
  - Foothills Research Center/CCT Research /ID# 260180, Phoenix, Arizona
  - Trialmed-Synexus Clinical Research US, Inc. - Tucson /ID# 258309, Tucson, Arizona
  - Preferred Research Partners /ID# 262786, Little Rock, Arkansas
  - Preferred Research Partners /ID# 273128, Little Rock, Arkansas
  - Hope Clinical Research /ID# 257867, Canoga Park, California
  - Axiom Research /ID# 257833, Colton, California
  - Neuro Pain Medical Center /ID# 257155, Fresno, California
  - Axiom Research, LLC-Los Angeles /ID# 264085, Glendale, California
  - Sun Valley Research Center /ID# 257152, Imperial, California
  - Axiom Research - Irvine /ID# 264083, Irvine, California
  - Collaborative Neuroscience Research CNS /ID# 257828, Los Alamitos, California
  - Los Angeles Headache Center /ID# 257237, Los Angeles, California
  - Pharmacology Research Institute (PRI) - Newport Beach (Wake) /ID# 257158, Newport Beach, California
  - Artemis Institute for Clinical Research - San Diego /ID# 257134, San Diego, California
  - M3 Wake Research - Convoy /ID# 257897, San Diego, California
  - Optimus Medical /ID# 257856, San Francisco, California
  - New England Institute for Clinical Research /ID# 264019, Stamford, Connecticut
  - Neurology Offices of South Florida, PLLC /ID# 257161, Boca Raton, Florida
  - Accel Research Sites Network - DeLand Clinical Research Unit /ID# 257403, DeLand, Florida
  - Indago Research & Health Center /ID# 277943, Hialeah, Florida
  - Accel Research Sites - Lakeland Clinical Research Unit /ID# 257874, Lakeland, Florida
  - Well Pharma Medical Research /ID# 257199, Miami, Florida
  - Sensible Healthcare /ID# 257198, Ocoee, Florida
  - Clinical Neuroscience Solutions, Inc /ID# 257190, Orlando, Florida
  - Conquest Research /ID# 258314, Winter Park, Florida
  - NeuroTrials Research /ID# 274507, Atlanta, Georgia
  - Clinical Research Atlanta - Headlands LLC /ID# 260181, Stockbridge, Georgia
  - Hawaii Pacific Neuroscience /ID# 274469, Honolulu, Hawaii
  - Velocity Clinical Research - Boise /ID# 257135, Meridian, Idaho
  - Healthcare Research Network /ID# 257868, Tinley Park, Illinois
  - Deaconess Midtown Hospital /ID# 257400, Evansville, Indiana
  - Accellacare - McFarland Clinic /ID# 257834, Ames, Iowa
  - Alliance for Multispecialty Research LLC /ID# 257839, Newton, Kansas
  - Collective Medical Research /ID# 257131, Overland Park, Kansas
  - Alliance for Multispecialty Research - Wichita East /ID# 257148, Wichita, Kansas
  - Tandem Clinical Research - Marrero - Barataria Boulevard /ID# 260146, Marrero, Louisiana
  - IMA Clinical Research Monroe - Wood /ID# 259362, Monroe, Louisiana
  - Headlands PharmaSite /ID# 257208, Baltimore, Maryland
  - Boston Clinical Trials /ID# 257132, Boston, Massachusetts
  - BTC of New Bedford /ID# 257128, New Bedford, Massachusetts
  - MedVadis Research /ID# 257156, Waltham, Massachusetts
  - Michigan Headache & Neurological Institute (MHNI) /ID# 257179, Ann Arbor, Michigan
  - Memorial Healthcare Institute For Neuroscience /ID# 274663, Owosso, Michigan
  - Proven Endpoints LLC /ID# 273796, Ridgeland, Mississippi
  - HealthCare Research Network - Hazelwood /ID# 257402, Hazelwood, Missouri
  - Clinvest Research LLC /ID# 257215, Springfield, Missouri
  - Methodist Physicians Clinic/CCT Research /ID# 260167, Fremont, Nebraska
  - Cognitive Clinical Trials (CCT) - Papillion /ID# 260174, Papillion, Nebraska
  - IMA Clinical Research Las Vegas /ID# 258679, Las Vegas, Nevada
  - Wr-Crcn, Llc /Id# 257895, Las Vegas, Nevada
  - Bio Behavioral Health, Inc /ID# 257140, Toms River, New Jersey
  - IMA Clinical Research Warren /ID# 263641, Warren Township, New Jersey
  - Albuquerque Clinical Trials, Inc. /ID# 257212, Albuquerque, New Mexico
  - Dent Neurologic Institute - Amherst /ID# 257219, Amherst, New York
  - IMA Clinical Research Westchester /ID# 259157, Hartsdale, New York
  - Fieve Clinical Research, Inc. /ID# 257177, New York, New York
  - Rochester Clinical Research /ID# 257193, New York, New York
  - True North Neurology /ID# 274672, Port Jefferson Station, New York
  - Upstate Clinical Research Associates /ID# 257163, Williamsville, New York
  - Headache Wellness Center /ID# 257136, Greensboro, North Carolina
  - Accellacare /ID# 257731, Winston-Salem, North Carolina
  - Accellacare /ID# 257850, Winston-Salem, North Carolina
  - Lillestol Research, LLC /ID# 257896, Fargo, North Dakota
  - CTI Clinical Research Center /ID# 257162, Cincinnati, Ohio
  - C7 Research /ID# 272815, Cleveland, Ohio
  - Centricity Research Columbus /ID# 257221, Columbus, Ohio
  - Wright State Physicians Health Center /ID# 274708, Fairborn, Ohio
  - Lynn Institute of Oklahoma City /ID# 257857, Oklahoma City, Oklahoma
  - Central States Research /ID# 277867, Tulsa, Oklahoma
  - Summit Research Network - Portland - Northwest Vaughn Street /ID# 257139, Portland, Oregon
  - Abington Neurological Associates - Abington /ID# 257164, Abington, Pennsylvania
  - Clinical Research of Philadelphia, LLC /ID# 257197, Philadelphia, Pennsylvania
  - Partners In Clinical Research /ID# 257855, Cumberland, Rhode Island
  - Premier Neurology /ID# 260359, Greenville, South Carolina
  - Coastal Carolina Research Center - North Charleston /ID# 257227, North Charleston, South Carolina
  - WR-ClinSearch /ID# 257160, Chattanooga, Tennessee
  - KCA Neurology /ID# 274495, Franklin, Tennessee
  - Alliance for Multispecialty Research - Knoxville /ID# 257846, Knoxville, Tennessee
  - FutureSearch Trials of Neurology /ID# 257186, Austin, Texas
  - FutureSearch Trials of Dallas, LP /ID# 257142, Dallas, Texas
  - Elevate Clinical - Seabrook /ID# 274679, Houston, Texas
  - Houston Clinical Research Associates /ID# 272077, Houston, Texas
  - Red Star Research, LLC /ID# 257871, Lake Jackson, Texas
  - Radiance Clinical Research /ID# 271727, Lampasas, Texas
  - Epic Clinical Research - Lewisville /ID# 274480, Lewisville, Texas
  - Sms Clinical Research /ID# 278443, Mesquite, Texas
  - Clinpoint Trials /ID# 274524, Waxahachie, Texas
  - Foothill Family Draper Clinic /ID# 277876, Draper, Utah
  - Advanced Research Institute /ID# 257853, Ogden, Utah
  - J. Lewis Research - Salt Lake City - Foothill Drive /ID# 277877, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South /ID# 258305, Salt Lake City, Utah
  - Highland Clinical Research /ID# 257137, Salt Lake City, Utah
  - Charlottesville Medical Research /ID# 257154, Charlottesville, Virginia
  - Alliance for Multispecialty Research - Clinical Research Associates /ID# 257851, Norfolk, Virginia
  - Northwest Clinical Research Center /ID# 257381, Bellevue, Washington
  - Puget Sound Neurology /ID# 257174, Tacoma, Washington
  - Vaught Neurological Services /ID# 267519, Beckley, West Virginia
  - West Virginia Univ School Med /ID# 258898, Morgantown, West Virginia
  - Mind+ Neurology /ID# 274486, Mequon, Wisconsin
- Puerto Rico (3):
  - ISIS Clinical Research Center /ID# 262858, Guaynabo
  - Instituto De Neurologia Dra. Ivonne Fraga, Psc /ID# 262852, San Juan
  - BDH Research /ID# 262851, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-714